CLINICAL TRIAL: NCT06233487
Title: Reliability of Ultrasound Metrics Used in Hip Dysplasia Diagnostics - a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Hans-Christen Husum, Postdoctoral Research Fellow, Department of Radiology, Principal Investigator, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-49-72-4-18
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Masking Description: The radiologist will be blinded to each others measurements, until all examinations have been performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double measurements (Other): All included children will have double measurements of the investigated ultrasound methodologies performed by two separate musculoskeletal radiologists.
  Interventions: Diagnostic Test: Repeat hip ultrasound measurements

INTERVENTIONS:
Diagnostic Test: Repeat hip ultrasound measurements — See earlier

SUMMARY:
Several measurements are used to evaluate hip dysplasia in hip ultrasound of children. Despite having being used since the 1980s, reliability studies have failed to find acceptable reliaiblity values for the gold standard ultrasound methods.

This study will evaluate three ultrasound measurement methodologies in a high quality controlled setting, to investigate the best achieveable reliability and agreement of the investigated measurements used in hip dysplasia diagnostics.

DETAILED DESCRIPTION:
In DDH diagnostics, measurements of acetabular alpha angles and femoral head coverages (FHC), developed by Graf and Harcke/Terjesen respectively, have been gold standard since the 1980s. Despite their widespread use, the reliability of these measurements has been questioned due to the relative complexity of acquiring the necessary corIDrect frontal 2D plane or "standard plane". In the only meta-analysis of the reliability of ultrasound (US) metrics in dysplasia, the interrater reliability of the alpha angles was mediocre while the reliability of the FHC was poor. Critics of these findings however argue that the low reliability reported in studies are due to misinterpretation and misapplication of the Graf method.

The pubo-femoral distance (PFD) was proposed in 2013 as a new measurement for assessing DDH, while the reliability is reportedly higher than the gold standard US methods, it has never been directly compared to these.

This study aims to evaluate the inter- and intrarater reliability of Graf's alpha and beta angles, the FHC and PFD in children referred for hip US in a selective ultrasound screening program for DDH.

ELIGIBILITY:
Inclusion Criteria:

* Children referred to the radiological outpatient at AUH for hip ultrasound examination, suspect of DDH.
* Children receiving follow-up ultrasound for previously diagnosed DDH

Exclusion Criteria:

* Children deemed too agitated to participate in hip US with double measurements by two radiologists.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-02-07 (Actual); Study Completion 2026-02-07 (Actual)

PRIMARY OUTCOMES:
Reliability and agreement in Alpha/Beta angles, Femoral head coverage and Pubo-femoral distance | Ultrasound measurements collected during the ultrasound examination by both radiologists
  For all included ultrasound measurement methods the following will be reported:
  Inter- and intrarater reliability will be evaluated using the intraclass correlation coefficient (ICC) and interpreted with ICC values between 0-0.5, 0.5-0.75, 0.75-0.9 and above 0.9 indicating poor, moderate, good and excellent reliability respectively.
  Agreement will be evaluated using Bland-Altman plots (to check for systematic bias) and mean absolute measurement differences between raters.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, analysis plan, and analytic code will be available upon written request to the first author.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study has been published (expected end 2024)
Access Criteria: upon written request to the first author.